CLINICAL TRIAL: NCT01243229
Title: Genetic Analysis of Congenital Diaphragmatic Disorders
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Luca Brunelli, M.D., University of Utah
Other Study IDs: 35848
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Congenital Diaphragmatic Hernia; Congenital Diaphragmatic Eventration; Congenital Hiatal Hernia; Congenital Diaphragmatic Disorders
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood or buccal swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to understand the genetic causes of congenital diaphragmatic disorders (CDD), namely congenital diaphragmatic hernia (CDH), eventration and hiatal hernia.

Specifically, the investigators plan to:

1. Ascertain informative families and sporadic cases with congenital diaphragmatic disorders and obtain appropriate phenotypic data and genetic material (peripheral blood and/or diaphragm tissue sample).
2. Localize the gene(s) for CDD to specific chromosomal segments using linkage analysis, and determine the role of somatic mutations in CDD.
3. Isolate and characterize genes involved in the pathogenesis of CDD.
4. Develop molecular markers that will facilitate accurate diagnosis (including prenatal diagnosis) and permit correlation of phenotypic variation with specific mutations.
5. Compare RNA-sequencing from tissue samples of children without CDH to those children with CDH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a congenital diaphragmatic disorder

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Newborns, children and adults affected by congenital disorders of the diaphragm, such as congenital diaphragmatic hernia, eventration and hiatal hernia.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2010-10; Primary Completion 2018-02-28 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Genes implicated in CDD can be identified by linkage analysis | 5 years
  Using the Utah Population Database, genes implicated in CDD can be identified by linkage analysis

SECONDARY OUTCOMES:
Develop molecular markers that will facilitate accurate diagnosis of CDD and CDH. | 5 years
  Develop molecular markers that will facilitate accurate diagnosis (including prenatal diagnosis) and permit correlation of phenotypic variation with specific mutations by localizing the gene(s) for CDH to specific chromosomal segments using linkage analysis in familial cases. In sporadic cases, characterize the role of somatic mutations in CDDs by using a candidate gene approach, and comparative genomic hybridization (CGH) arrays.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Brunelli, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University Hospital, Salt Lake City, Utah